CLINICAL TRIAL: NCT05938699
Title: Aqueous Humor Dynamics of NCX 470 Ophthalmic Solution - A Double-Masked, Placebo-Controlled, Phase 3b Clinical Trial (Whistler)
Brief Title: Aqueous Humor Dynamics of NCX 470 Ophthalmic Solution
Acronym: Whistler
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NCX 470-05
Record Dates: First submitted 2023-06-15; First posted 2023-07-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Open Angle Glaucoma
Keywords: glaucoma; NCX 470; nitric oxide; prostaglandin analogue
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Nitric Oxide; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NCX 470 0.1% (Active Comparator): NCX 470 0.1% - one drop in the randomized eye once a day for 8 days
  Interventions: Drug: NCX 470
- Placebo (Placebo Comparator): Artificial tears - one drop in the randomized eye once a day for 8 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NCX 470 — NCX 470 0.1% vs Placebo
  Other Names: nitric oxide (NO)-donating bimatoprost prostaglandin analog
  Arms: NCX 470 0.1%
Drug: Placebo — NCX 0.1% vs Placebo
  Other Names: Artificial tears
  Arms: Placebo

SUMMARY:
This is a double-masked, placebo-controlled study which will determine the action of NCX 470 ophthalmic solution, 0.1% on aqueous humor dynamic parameters in healthy volunteers or subjects with OHT.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Either gender
3. Subjects without glaucoma
4. Qualifying IOP at Screening Visit

Exclusion Criteria:

1. Narrow anterior chamber angles or disqualifying central corneal thickness in either eye
2. Clinically significant ocular disease in either eye
3. Uncontrolled systemic disease
4. Serious hypersensitivity to topical anesthetic eye drops
5. Subjects with a known hypersensitivity or contraindications to any of the ingredients in the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Change in AHD | 8 days
  The primary efficacy endpoint is change from baseline in aqueous humor dynamics AHD). AHD is calculated by using well establish techniques which include capturing the following:
  Aqueous humor flow rates from fluorescein clearance; Outflow facility using constant weigh tonography; Episcleral venous pressure using a venomanometer.
  The change in ADH will be calculate in normals following 8 (±1) days of dosing of NCX 470 0.1% compared to placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No